CLINICAL TRIAL: NCT05796895
Title: Development and Testing of a Videogame Intervention for Improving the Health-related Quality of Life (HrQOL) of Children With Cancer
Brief Title: A Videogame Intervention for Children With Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Sehrish Sajjad, Principal Investigator, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-6833-21251
Record Dates: First submitted 2023-02-23; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Cancer
Keywords: Childhood cancer; Videogame; Health-related Quality of Life; Mixed Methods; Low and Middle-Income Country
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: There will be two groups in parallel. The first will be the intervention group in which children will be provided with the videogame intervention for eight weeks. Children will play the videogame and learn about symptom management strategies through the game tasks. The children will complete the tasks, score points, and progress to the next game. The videogame will be connected to a web-based portal through which the research team will retrieve data regarding the progress of the children's gameplay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Children will be provided with the videogame through which we will teach them symptom management strategies.
  Interventions: Behavioral: Videogame
- Attention Control Group (Active Comparator): An attention control group will be used in this study for comparison with the intervention group. Children of the attention control group will receive weekly WhatsApp messages on general health behaviours.
  Interventions: Behavioral: WhatsApp

INTERVENTIONS:
Behavioral: Videogame — Children will be provided with the videogame for eight weeks, through which they will be taught symptom management strategies. Children and their parents will be telephoned every week by a nurse to inquire whether children performed the strategies taught to them and if they have any health concerns. Children and parents can also call the nurse educator if they have any questions. Their queries/concerns will be responded to by the nurse educator in consultation with the clinical health experts (doctors and nurses) in the research team.
  Arms: Intervention Group
Behavioral: WhatsApp — Children will be provided with weekly WhatsApp messages on healthy behaviors. Children and their parents will be telephoned every week by a nurse to inquire whether they have any health concerns. Children and parents can also call the nurse educator if they have any questions. Their queries/concerns will be responded to by the nurse educator in consultation with the clinical health experts (doctors and nurses) in the research team.
  Arms: Attention Control Group

SUMMARY:
The investigators aim to improve the quality of life and well-being of children with cancer in low- and middle-income countries through a videogame intervention. In this study, first, the investigators will identify common symptoms faced by children with cancer during their cancer treatment and their parents. Based on what they share, the investigators will develop a videogame to teach children how to manage their symptoms at home. The investigators will provide the videogame intervention to a group of children with cancer, and the other group will receive general Whatsapp messages to improve their overall health. Through survey questions, the investigators will test the videogame intervention from the first group of children to see whether their symptom distress decreased and their quality of life improved. The investigators will also test the videogame intervention for its usefulness, through interviews from children, their parents, and healthcare providers.

DETAILED DESCRIPTION:
The prevalence of childhood malignancies has been rising worldwide. Chemotherapy and radiation cause severe side effects harming children's health-related quality of life (HRQOL) and causing symptom distress. Children who actively participate in their self-care make healthier choices for themselves. Several studies suggest that children engage better with digital health interventions (DHIs) and learn self-care quickly, consequently improving their health outcomes. Videogames are an example of evolving DHI to engage children and educate them about symptom management.

An exploratory sequential mixed methods design will be employed. In the first phase, the investigators conducted in-depth interviews with child-parent dyads to explore their experiences with cancer treatment and their preferences regarding the videogame's design. In the study's second phase, the investigators will work with clinical and digital health professionals to design the videogame based on the interview results. The investigators will conduct a Randomized Controlled Pilot and Feasibility Study (Pilot-RCT) in the third phase. The investigators will provide the intervention group's children access to a gaming application to teach children how to take care of themselves and manage symptoms associated with cancer treatment. Weekly WhatsApp messages on healthy behaviours will be sent to children in the attention control group.

ELIGIBILITY:
Inclusion Criteria:

* 8-18 years old
* Diagnosed with any type and stage of cancer within six months of the diagnosis.
* Receiving active treatment
* Can comprehend Urdu and/or English language
* Have access to an android smartphone/tablet for at least 30 minutes/day to play the video game (either they or their parents own a smartphone)
* Provide informed assent and their parents provide written permission/consent.

Exclusion Criteria:

* Severely or critically ill
* Admitted only for blood transfusion without a diagnosis of cancer
* Receiving palliative treatment.
* Have presence of any diagnosed sight, hearing, cognitive impairment, or upper limb deformity limiting them to play the videogame.
* If already playing any videogame having the same content

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Determine change in the Health-related Quality of Life (HRQOL) between study groups, from baseline at eight weeks, on the Pediatric Quality of Life Inventory Generic Core Scale (PedsQL 4.0). | Baseline, pre-intervention and eight weeks post-intervention
  Children of both groups will be administered the Pediatric Quality of Life Inventory Generic Core Scale (PedsQL 4.0) at baseline and at eight weeks to assess the change in the Health-related Quality of Life (HRQOL). The responses on individual items are recorded on a 5-point Likert scale (0 = never a problem to 4 = almost always a problem), and the scores are converted from 0 to 100. The higher the score, the more favorable is the HrQOL.
Determine change in the Health-related Quality of Life (HRQOL) between study groups, from baseline at eight weeks, on the Pediatric Quality of Life Inventory Cancer Module (PedsQL 3.0). | Baseline, pre-intervention and eight weeks post-intervention
  Children of both groups will be administered the Pediatric Quality of Life Inventory Cancer Module (PedsQL 3.0) at baseline and at eight weeks to assess the change in the Health-related Quality of Life (HRQOL).The responses on individual items are recorded on a 5-point Likert scale (0 = never a problem to 4 = almost always a problem), and the scores are converted from 0 to 100. The higher the score, the more favorable is the HrQOL.

SECONDARY OUTCOMES:
Determine change in the Cancer Symptoms Frequency and Distress between study groups, from baseline at eight weeks, on the Memorial Symptom Assessment Scale Short Form (MSAS-SF). | Baseline, pre-intervention and eight weeks post-intervention
  Children of both groups will be administered the Memorial Symptoms Assessment Scale Short Form at baseline and at eight weeks to assess the change in the symptom frequency and distress. They will be asked to report the frequency (i.e. rarely, occasionally, frequently, almost constantly) and distress (not at all, a little bit, somewhat, quite a bit, very much) of each symptom. (Higher score indicates more distress and frequency).

OTHER OUTCOMES:
Patient-reported Acceptability and Satisfaction of the videogame intervention on the Acceptability E-scale. | Eight weeks post-intervention
  Children of the intervention group will be administered Acceptability E-scale to assess the acceptability and satisfaction of the videogame intervention, on a Likert scale of 1 (very unacceptable and dissatisfying) to 5 (very acceptable and very satisfying).
Patient-reported Appropriateness of the videogame intervention assessed in qualitative interviews from the intervention group child-parent dyads. | Eight weeks post-intervention
  The intervention group child-parent dyads will be interviewed qualitatively eight weeks after the intervention to share their experience with the videogame intervention. Questions will be asked from them to explore appropriateness of the videogame intervention. Similarly doctors and nurses from the oncology setting will be inquired about the appropriateness of the videogame intervention in a focus group discussion.
Cost of development of the videogame intervention as determined from the videogame development team. | Baseline, pre-intervention
  The videogame development cost will be reported in Pakistani rupees.
Proportions of children recruited, refused to participate, and loss to follow-up along with their reasons of refusal to participate and loss to follow-up. | Eight weeks post-intervention
  Proportions of children recruited, refused to participate, and loss to follow-up along with their reasons for refusal to participate and loss to follow-up in both groups will be reported, which will indicate the feasibility of the study.
Total game score obtained by the participants in the videogame. | Eight weeks post-intervention
  The intervention group children's progress of the videogame as assessed via the total game score obtained will be reported.

IPD SHARING:
Plan to Share IPD: No
Data obtained through this study will be deidentified and findings will be shared in an aggregated form in the reports and publications.

REFERENCES:
- [Derived] Sajjad S, Gul RB, Sayani S, Fadoo Z, Abbasi AN, Barolia R. Development and testing of a videogame intervention for symptom management among 8-18 years old children with cancer: a study protocol. BMJ Paediatr Open. 2024 Oct 16;8(1):e002679. doi: 10.1136/bmjpo-2024-002679. PMID 39414341